CLINICAL TRIAL: NCT05643027
Title: A Novel Intervention for Avoidance-Related Opioid Misuse in Patients With Cancer
Brief Title: A Novel Intervention for Patients With Cancer
Acronym: ACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Miryam Yusufov, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-587; 1K08CA259538-01A1 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-12-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Substance Use; Cancer; Psychological
Keywords: feasibility; acceptability
MeSH Terms: conditions — Substance-Related Disorders; Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INTERVENTION FOR AVOIDANCE-RELATED OPIOID MISUSE (Other): Participants will participate in a six-session behavioral intervention, delivered by a licensed clinical psychologist.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Six-session, skills-based behavioral intervention targeting risk factors for opioid use disorder in the context of cancer

SUMMARY:
This research study is being done to develop an intervention for psychological symptoms that patients diagnosed with cancer may experience. Psychological symptoms may include thoughts, feelings, emotions, and memories

The names of the study intervention and research activities involved in this study are/is:

* Acceptance & Commitment Therapy (ACT) for Cancer (involving 6 sessions with a licensed clinical psychologist)
* Questionnaires
* Post-study interview

Consistent with the NIH Stage Model for Behavioral Intervention Development, the investigators have adapted an existing, empirically-validated intervention, Acceptance and Commitment Therapy (ACT), to address substance use disorder risk during cancer care. The core components of ACT are particularly well-suited to address the psychological processes underlying opioid misuse in individuals treated for cancer pain. The overarching aim is to assess the feasibility and acceptability of the intervention by conducting a randomized pilot trial of the revised intervention ("ACTION") for cancer patients on opioid therapy, and at risk for SUD.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first-time investigators are examining this psychological intervention in patients with cancer who are prescribed opioids and are receiving palliative care. This study is being conducted to develop a psychological intervention designed specifically for individuals with cancer. The purpose of this study is to determine how practical this intervention is, to determine patient satisfaction, and test the study procedures. The aims are to:

1. determine whether this intervention will be appropriate for further testing;
2. identify which parts of the protocol and procedures need to be modified; and
3. assess patients' reactions to this intervention.

This research study involves a psychological intervention for thoughts, feelings, emotions, and memories that individuals diagnosed with cancer may have.

The names of the study intervention and research activities involved in this study are/is:

* Acceptance & Commitment Therapy (ACT) for Cancer (involving 6 sessions with a licensed clinical psychologist)
* Questionnaires
* Post-study interview

The research study procedures include: screening for eligibility and study treatment including evaluations, 6 visits, and a post-study interview.

Participants will be on this research study for up to 2 months.

It is expected that about 10 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* have an estimated survival time of at least 6 months (as estimated by palliative care provider)
* score at least 4 on the Opioid Risk Tool (ORT)
* have been diagnosed with any cancer, including hematologic malignancies
* performance status criterion of 0, 1, or 2 [ with 0 indicating that the patient is asymptomatic, 1 that the patient is symptomatic but fully ambulatory, and 2 that the patient is symptomatic and in bed <50% of the day]

Exclusion Criteria:

* Patients with a score at least 3 to ensure that all enrolled patients are able to participate in the intervention, complete assessments, ensure that no patients who are too sick to participate are enrolled; this will enhance the rigor of the study)
* currently be on opioid therapy
* not meet criteria for current substance use disorder
* assessed by the Diagnostic & Statistical Manual of mental disorders; DSM-5 or be receiving substance use disorder treatment; and speak and comprehend English sufficiently to be able to participate in psychotherapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention, defined as an enrollment rate of at least 60% | 1 year
  enrollment rate of at least 60% and retention rate of at least 75%
Acceptability of the intervention, measured by Client Satisfaction Questionnaire (CSQ-8) scores | 1 year
  Acceptability of the intervention, measured by CSQ-8 scores and patient reported feedback during exit interviews. On the CSQ-8, some items are reverse scored but higher scores mean greater satisfaction. Min value = 8, max value = 32

SECONDARY OUTCOMES:
Depression, measured by the Patient Health Questionnaire (PHQ-9) | 1 year
  patient reported depression symptoms, as measured by the PHQ-9; higher scores represent a worse outcome (i.e., more depression); min value = 1; max value = 27
anxiety, as measured by the Generalized Anxiety Disorder questionnaire (GAD-7) | 1 year
  anxiety, as measured by the GAD-7; higher scores indicate a worse outcome (i.e., greater anxiety); min value = 0; max value = 21
opioid misuse behaviors and consequences, as measured by the Current Opioid Misuse Measure (COMM) | 1 year
  opioid misuse behaviors and consequences, as measured by the COMM; with a sum of questions that is less than 9 reflecting no misuse and greater or equal to 9 reflecting misuse

CONTACTS AND LOCATIONS:
Overall Officials: Miryam Yusufov, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Yusufov M, Pirl WF, Greer JA, Mazzola E, Dalrymple KL, Tulsky JA, Braun IM, McHugh RK. Study protocol for a pilot randomised controlled trial of a virtually delivered behavioural intervention (ACTION) for adults with cancer at risk for opioid use disorder. BMJ Open. 2024 Dec 5;14(12):e096546. doi: 10.1136/bmjopen-2024-096546. PMID 39638585